CLINICAL TRIAL: NCT06358287
Title: Neural Correlates of Auriculotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keith M. Vogt, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Keith M. Vogt, MD, PhD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030375
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cryogenic Auriculotherapy Treatment (Experimental): Compressed nitrogen is used to create a 'cryogenic needle', using a cryopunctor device. An orifice is placed in appropriate acupoint and nitrogen flow is used to cool and activate the point. This will occur on each ear with the following points being targeted: Omega 2, Omega, spine location point, and 3 points of the pain pathway including the sensory master point (SMP), the master point of the reticule (MPR), and the thalamus (T) as well as the corpus callosum (CC) point, the amygdala, rhinencephalon, hippocampus, FSHLH, ACTH, anterior and posterior white commissure points, and the corresponding sympathetic sensory and motor nerve points.
  Interventions: Procedure: cryogenic auriculotherapy

INTERVENTIONS:
Procedure: cryogenic auriculotherapy — Compressed nitrogen is used to create a 'cryonic needle', using a cryopunctor device. An orifice is placed in appropriate acupoint and nitrogen flow is used to cool and activate the point.

SUMMARY:
Chronic pain continues to be a major health issue, creating a significant societal burden, as it is an independent risk factor for opioid use disorder (OUD) and deaths. Acute pain episodes can often engender OUD due to lack of effective strategies to treat pain and prevent the transition to chronic pain. One potential non-opioid method for pain relief is auriculotherapy (AT), where acupuncture-like treatment is administered to the ear. The objective of this pilot study is to illustrate that AT-related brain effects can be found using functional connectivity MRI (fcMRI) in patients with low back pain.

DETAILED DESCRIPTION:
Chronic pain continues to be a major health issue, creating a significant societal burden, as it is an independent risk factor for opioid use disorder (OUD) and deaths. Acute pain episodes can often engender OUD due to lack of effective strategies to treat pain and prevent the transition to chronic pain. One potential non-opioid method for pain relief is auriculotherapy (AT), where acupuncture-like treatment is administered to the ear. This technique has recently been applied, with analgesia lasting for weeks, to patients with acute peri-operative pain at Shadyside hospital, but the mechanism of action of AT remains unclear.

Our overall objective is the determine the mechanism that drives AT-induced pain relief and utilize this tool as an adjuvant in our efforts to reduce the nation's reliance on opioids for pain relief. The objective of this pilot study is to illustrate that AT-related brain effects can be found with functional MRI (fMRI) for low back pain, with which the investigators have much experience. Our hypothesis is that AT reduces pain score and the abnormal brain connectivity associated with low back pain. This will identify areas of brain activity that correlate with symptom improvement after AT, allow hypothesis generation for further testing, and provide the data necessary for power calculations for an appropriately powered study in subsequent NIH HEAL grant applications.

Aim 1. Identify brain activity changes after treatment with AT. The investigators previously characterized the resting state brain activity in patients with chronic low back pain and identified key brain areas with connectivity changes related to pain state. Guided by that study, the investigators will determine if AT causes changes in resting state brain activity by comparing scans acquired before and after AT. Specifically, connectivity between the default mode network (DMN) and the insula and anterior cingulate cortex (ACC) will be examined. Changes in these areas will support the theory that AT's modulation of neural processing can be objectively measured and further characterized in a larger study.

Aim 2. Determine if detailed psychometric pain assessments demonstrate changes across AT therapy. Detailed information regarding the change in pain scores after AT are not available. Patients will complete the Patient-Reported Outcome Measurement Information System (PROMIS) Questionnaire-29 and the global impression of change questionnaires, among others, prior to and after AT treatment. This aim will also illustrate expertise in AT for chronic conditions, complimenting current efforts to demonstrate the same in acute pain after shoulder surgery. The combination of this data with the on-going acute pain study will provide the preliminary psychometric data necessary to support future NIH funding.

Aim 3. Gain insight into whether placebo mechanisms play a role in AT's efficacy. Complimentary medicine treatments such as AT are often suggested to work via placebo mechanisms. Recent work suggests that the connectivity of the right midfrontal gyrus (r-MFG) predicts the response to placebo therapy. The investigators will correlate the pain score response to AT treatment with r-MFG connectivity to determine if greater pain reduction is seen in those with greater r-MFG activity, suggesting overlap with circuits underlying placebo analgesia.

Aim 4. A small aliquot of blood will be obtained and markers of inflammation will be assessed using an ultrasensitive human 10-plex panel, which quantifies circulating levels of tumor necrosis factor (TNF-α), Interleukin (IL)-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, Interferon-y (IFNγ), and cytokine, granulocyte macrophage-colony stimulating factor (GM-CSF).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above.
* Experiencing low back pain for > 1 month and seeking treatment.
* Literate for reading and writing in English, decision competent, willing and able to provide written informed consent, and able to complete the study's schedule of assessments.

Exclusion Criteria:

* Subjects under 18 years of age.
* History of claustrophobia.
* Having non-MRI safe metallic or foreign objects in their body.
* History of dementia.
* History of sensory or motor deficits that preclude participation in pain fMRI.
* History of clinically unstable systemic illness that is judged to interfere with the study.
* Pregnancy or the intent to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Default Mode Network (DMN)-to-Anterior Cingulate Cortex (ACC) connectivity | Day 3 of participation
  Group average difference in connectivity will be calculated as pre-treatment vs. post-treatment statistical contrasts. Connectivity change will have a threshold at the connection level with p < 0.001. In this framework, a positive T-Score indicates greater connectivity before treatment (a decrease in connectivity after treatment).

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) Severity Scores MRI #1 | Day 3 of participation
  The Brief Pain Inventory Pain Severity is based on a scale of 0= no pain at all, and 10= the worst pain imaginable. This outcome measurement is recorded as mean(SD).
BPI Pain Severity Scores MRI #2 | Day 3 of participation
  The Brief Pain Inventory Pain Severity is based on a scale of 0= no pain at all, and 10= the worst pain imaginable. This outcome measurement is recorded as mean(SD).
General Anxiety Disorder-7 (GAD-7) Scoring | Day 3 of participation
  The General Anxiety Disorder-7 has a minimum score of 0, and a maximum score of 21. The average score will be recorded as mean(SD).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Vogt, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Montefiore, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share this preliminary data.